CLINICAL TRIAL: NCT02843139
Title: Circulating microRNAs as Novel Prognostic Biomarkers in Obese Preschoolers at Risk for Type 2 Diabetes in Adulthood
Brief Title: Circulating microRNAs for Discriminating Obese Preschoolers at Risk of Diabetes
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Vice-president, Nanjing Medical University
Other Study IDs: NMU-201487
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Discriminate Obese Children at Risk for Diabetes.
Keywords: Circulating microRNA; Childhood obesity; Adulthood diabetes
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children group: Children recruiters were categorized into three groups: obesity, overweight and normal control based on World Health Organization child growth standards.
- Adults group: Adults with type 2 diabetes were defined if the individual had a fasting plasma glucose (FPG) level ≥ 7.0 mmol/L.

SUMMARY:
Childhood obesity certainly increases susceptibility to type 2 diabetes (T2D) in adulthood. Recently, microRNAs (miRNAs) are closely related to various diseases and have been suggested as valuable biomarkers. Here, we sought to identify potential miRNAs to discriminate obese children at risk for diabetes in future.

DETAILED DESCRIPTION:
This study was designed to screen the circulating miRNAs in association with progression from children obesity to type 2 diabetes (T2D) in adulthood. Serum samples were evaluated in a 3 step procedure: 1) discovery study, in which samples from obese children and healthy controls were pooled for miRNA sequecing experiment; 2) cross-sectional validation study, in which miRNAs of interest were validated in all individuals (obese children, overweight children and normal controls); 3) longitudinal validation study, in which the candidate miRNAs were estimated in newly diagnosed diabetes patients and normal glucose tolerance controls (NGT). The final determined miRNAs were further confirmed though primary function studies.

ELIGIBILITY:
Inclusion Criteria:

Obese preschoolers; Adults with type 2 diabetes; Age-matched healthy controls.

Exclusion Criteria:

-

Ages: 48 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children recruiters were categorized into three groups: obesity, overweight and normal control based on World Health Organization child growth standards. Adults with type 2 diabetes were defined if the individual had a fasting plasma glucose (FPG) level ≥ 7.0 mmol/L.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
It is expected that the identification of circulating miRNAs as potential biomarkers may facilitate to the diagnosis of obese preschoolers at high risk for developing diabetes. | 50-70 month old

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Maternal and Child Health Care Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided